CLINICAL TRIAL: NCT05197920
Title: Diabetes RElated to Acute Pancreatitis and Its Mechanisms (DREAM) An Observational Cohort Study From the Type 1 Diabetes in Acute Pancreatitis Consortium (T1DAPC)
Brief Title: Diabetes RElated to Acute Pancreatitis and Its Mechanisms
Acronym: DREAM
Status: Recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Benaroya Research Institute (Other); Cedars-Sinai Medical Center (Other); University of Southern California (Other); Indiana University (Other); Johns Hopkins University (Other); Ohio State University (Other); Stanford University (Other); University of Florida (Other); AdventHealth (Other); University of Illinois at Chicago (Other); Northwestern University (Other); University of Minnesota (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Vernon Michael Chinchilli, Distinguished Professor, Milton S. Hershey Medical Center
Other Study IDs: Penn State College of Medicine; U01DK127384 (NIH)
Record Dates: First submitted 2021-12-11; First posted 2022-01-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Acute Pancreatitis
Keywords: Diabetes
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood (fasting blood glucose, islet autoantibodies, creatinine, complete blood count (CBC), RNAseq), stool (fecal elastase)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overriding objective of DREAM is to conduct a prospective longitudinal (36 months) observational clinical study to investigate the incidence, etiology, and pathophysiology of diabetes mellitus (DM) following acute pancreatitis (AP).

DETAILED DESCRIPTION:
The DREAM investigators will conduct dynamic metabolic testing that includes oral glucose tolerance testing (OGTT), mixed meal tolerance testing (MMTT), and frequently sampled intravenous glucose tolerance testing (FSIGTT). These tests will increase the sensitivity for DM diagnosis (with OGTT) and to assess beta cell function and other pancreatic and enteroendocrine hormones involved in maintaining glucose homeostasis (OGTT, MMTT and FSIGTT). The DREAM research hypotheses are as follows.

1. There is a cumulative increase in the risk of any type of DM after an episode of AP, and the development of DM after AP is influenced by several patient and disease-related factors (e.g. age, etiology, disease severity).
2. After AP is clinically resolved, there is ongoing subclinical beta cell damage that predisposes to delayed-onset of DM.
3. AP triggers an altered immune state in a subset of individuals that predisposes to islet autoimmunity and DM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pancreatitis (AP) 0-90 days prior to enrollment date
* Participant fully understands and is able to participate in all aspects of the study, including providing informed consent, completion of case report forms (CRFs), telephone interviews, metabolic testing, and planned longitudinal follow-ups

Exclusion Criteria:

* Diagnosis of definite chronic pancreatitis (CP) at enrollment based on either of the following criteria met by computed tomography (CT) scan (including non-contrast enhanced) or Magnetic resonance Imaging (MRI) or Magnetic Resonance Cholangiopancreatography (MRCP): (a) Parenchymal or ductal calcifications on CT scan (after excluding the possibility that calcifications are vascular); (b) Intraductal filling defects suggestive of calcifications on MRI and/or MRCP
* Potential participants with post-endoscopic retrograde cholangiopancreatography (post- ERCP) AP who are hospitalized for <48 hours.
* Prior (i.e., before enrollment) direct endoscopic necrosectomy of the pancreas or percutaneous necrosectomy or drainage of necrotic collection(s). Participants who require this during follow-up will remain in the study
* Pancreatic tumors, including ductal adenocarcinoma, neuroendocrine tumors, and metastasis
* Confirmed or suspected cystic tumor associated with main pancreatic duct dilation, or believed to be the cause of AP (in the site-PI's judgement)
* Prior pancreatic surgery, including, but not limited to: distal pancreatectomy, pancreaticoduodenectomy, pancreatic necrosectomy, Frey procedure
* Use of disallowed concomitant medications within 30 days prior to enrollment. A comprehensive list of disallowed medications will be included and routinely updated in the study's Manual of Procedures
* Severe systemic illness that in the judgement of the investigative team will confound outcome assessments of DM and immunological outcomes or pose additional risk for harms, including: history of solid organ transplant, acquired immunodeficiency syndrome (AIDS), active treatment for cancer (except non-melanoma skin cancer) within 12 months prior to enrollment, chronic kidney disease with estimate glomerular filtration rate (eGFR) < 30 or on dialysis prior to AP, and cirrhosis (based on imaging or biopsy), or any other medical condition that in the opinion of the site-PI carries a life expectancy of <12 months.
* Known pregnancy at the time of enrollment. Participants who become pregnant during follow-up will remain in the study, but may have modified study assessments for safety
* Incarceration
* Any other condition or factor that would compromise the participant's safety or the scientific integrity of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
diabetes mellitus (DM) following a qualifying episode of acute pancreatitis (AP) | any time during the 36-month longitudinal follow-up period
  time to onset of DM during the 36-month longitudinal follow-up period

SECONDARY OUTCOMES:
PROMIS Global Health | months 3, 12, 24, and 36
  Patient Reported Outcomes Measurement Information System (PROMIS) Global Health, converted to a t-score with a mean of 50 and a standard deviation of 10
PROMIS Pain Intensity | months 3, 12, 24, and 36
  Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity, measured on an 11-point scale from 0 (no pain ) to 10 (worst pain imaginable)
PROMIS-29 Physical Function | months 3, 12, 24, and 36
  PROMIS-29 Physical Function, converted to a t-score with a mean of 50 and a standard deviation of 10
PROMIS-29 Anxiety | months 3, 12, 24, and 36
  PROMIS-29 Anxiety, converted to a t-score with a mean of 50 and a standard deviation of 10
PROMIS-29 Depression | months 3, 12, 24, and 36
  PROMIS-29 Depression, converted to a t-score with a mean of 50 and a standard deviation of 10
PROMIS-29 Fatigue | months 3, 12, 24, and 36
  PROMIS-29 Fatigue, converted to a t-score with a mean of 50 and a standard deviation of 10
PROMIS-29 Sleep Disturbance | months 3, 12, 24, and 36
  PROMIS-29 Sleep Disturbance, converted to a t-score with a mean of 50 and a standard deviation of 10
PROMIS-29 Ability to Participate in Social Roles and Activities | months 3, 12, 24, and 36
  PROMIS-29 Ability to Participate in Social Roles and Activities, converted to a t-score with a mean of 50 and a standard deviation of 10
PROMIS-29 Pain Interference | months 3, 12, 24, and 36
  PROMIS-29 Pain Interference, converted to a t-score with a mean of 50 and a standard deviation of 10
OGTT Insulin Secretion | months 3, 12, 24, and 36
  Oral Glucose Tolerance Testing (OGTT) Insulin Secretion, as measured by the insulin area under the curve relative to the glucose area under the curve
OGTT Insulin Sensitivity Index | months 3, 12, 24, and 36
  Oral Glucose Tolerance Testing (OGTT) Insulin Sensitivity Index, as measured by the glucose disposal rate divided by the average plasma insulin concentration
MMTT Incretin Hormones: GIP and GLP-1 | months 3, 12, 24, and 36
  Mixed Meal Tolerance Testing (MMTT) Incretin Hormones: Glucose-dependent Insulinotropic Polypeptide (GIP, pmol/L) and Glucagon-like Peptide-1 (GLP-1, pmol/L)
MMTT Glucagon | months 3, 12, 24, and 36
  Mixed Meal Tolerance Testing (MMTT) Glucagon (pg/mL)
MMTT Pancreatic Polypeptide (PP) | months 3, 12, 24, and 36
  Mixed Meal Tolerance Testing (MMTT) Pancreatic Polypeptide (PP, pg/mL)
FSIGTT Acute Insulin Response to Glucose (AIRglu) | months 3 and 12
  Frequently Sampled Intravenous Glucose Tolerance Testing (FSIGTT) Acute Insulin Response to Glucose (AIRglu)
FSIGTT Acute C-peptide Response to Glucose (ACRglu) | months 3 and 12
  Frequently Sampled Intravenous Glucose Tolerance Testing (FSIGTT) Acute C-peptide Response to Glucose (ACRglu)
FSIGTT Total Body Insulin Sensitivity Index (SI) | months 3 and 12
  Frequently Sampled Intravenous Glucose Tolerance Testing (FSIGTT) Total Body Insulin Sensitivity Index (SI)
FSIGTT Total Body Insulin Sensitivity Index (SI) Disposition Index | months 3 and 12
  Frequently Sampled Intravenous Glucose Tolerance Testing (FSIGTT) Disposition Index (DI), calculated as the product of the AIRglu and the Total Body Insulin SI
Islet Autoantibodies | months 3, 12, 24, and 36
  Islet Autoantibodies
Fecal Elastase | months 3, 12, 24, and 36
  Fecal Elastase (ug/g)

CONTACTS AND LOCATIONS:
Overall Officials: Vernon M Chinchilli, PhD, Principal Investigator — Penn State College of Medicine; Dhiraj Yadav, MD, MPH, Study Chair — University of Pittsburgh; Melena D Bellin, MD, Study Chair — University of Minnesota; Phillip A Hart, MD, Study Chair — Ohio State University
Locations (13):
- United States (13):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - AdventHealth, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data from final locked datasets will be made available to other researchers outside the DREAM investigative team. The plan for data sharing incorporates a strategy that recognizes the importance of protecting participants' rights to individual privacy and is compliant with HIPAA regulations and NIH requirements (https://grants.nih.gov/grants/policy/data_sharing/).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available one year after publication of the primary manuscript of the DREAM study. The data will be available indefinitely at the NIDDK Central Repository.
Access Criteria: Instructions for requesting data from the NIDDK Central Repository appear at the following web site:
  https://repository.niddk.nih.gov/pages/overall_instructions/
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- See also: Public web site for the Type 1 Diabetes in Acute Pancreatitis Consortium — http://t1dapc.net